CLINICAL TRIAL: NCT00419133
Title: Immune Responses Following One Versus Two Doses of Killed Oral Cholera Vaccine in Eastern Kolkata, West Bengal, India
Brief Title: Immunogenicity of One Versus Two Doses of Killed Oral Cholera Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: National Institute of Cholera and Enteric Diseases, India (Other); Shantha Biotechnics Limited (Industry)
Responsible Party: Director General, International Vaccine Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C-8IR
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Cholera; Diarrhea; Vibrio Infections
Keywords: Cholera; Vaccine; Kolkata; West Bengal; India; Immunogenicity; Safety
MeSH Terms: conditions — Cholera; Diarrhea; Vibrio Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cholera Vaccine
  Interventions: Biological: Killed bivalent whole cell oral cholera vaccine
- 2 (Placebo Comparator): Placebo
  Interventions: Biological: Heat Killed E. coli Placebo

INTERVENTIONS:
Biological: Killed bivalent whole cell oral cholera vaccine — Each 1.5 mL dose, given orally, contains:
  V. cholerae O1 Inaba El Tor strain Phil 6973 formalin killed, 600 Elisa units (EU) LPS V. cholerae O1 Ogawa classical strain Cairo 50 heat killed 300 EU LPS V. cholerae O1 Ogawa classical strain Cairo 50 formalin killed 300 EU LPS V. cholerae O1 Inaba classical strain Cairo 48 heat killed 300 EU LPS V. cholerae O139 strain 4260B formalin killed 600 EU LPS
  Arms: 1
Biological: Heat Killed E. coli Placebo — Heat Killed E.coli in an optical turbidity identical to cholera vaccine, given in a 1.5 mL oral dose.
  Arms: 2

SUMMARY:
The purpose of this study is to compare the safety and immunogenicity of one and two doses of the killed oral cholera vaccine.

DETAILED DESCRIPTION:
Cholera is an important public health problem worldwide, particularly in endemic areas of the developing world. In 2004, 101 383 cholera cases and 2345 deaths were reported to the WHO. Provision of safe water and food, adequate sanitation and improved personal and community hygiene are the main public health interventions against cholera. These measures cannot be implemented in the near future in the most cholera-endemic areas.

Phase II trials of this reformulated killed oral cholera vaccine were performed in SonLa, Vietnam and Kolkata, India. Significant vibriocidal antibody responses were observed among vaccine recipients.

Distribution of 2 doses of the cholera vaccine is often difficult in field settings and limits its utility in emergency situations, since an interval of 2 weeks is usually required between doses. Recent data from Vietnam suggests that greater vibriocidal responses following 2 doses are elicited compared to previous formulations. Furthermore, in a study in Bangladesh comparing immune responses to the vaccine among children supplemented with vitamin A and zinc, seroconversion after the first dose was robust in all groups suggesting that one dose may be used in the control of cholera.

Data regarding the immune response following one dose of this reformulated vaccine is currently unavailable. If a single dose of this vaccine is confirmed to be immunogenic to recipients, then this vaccine may be used more extensively for public health purposes, especially during times of outbreaks.

The objective of this study is to confirm the safety of the killed oral cholera vaccine among adult and children volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and non-pregnant female adults aged 18-40 years and healthy children aged 1-17 years

All subjects must satisfy the following criteria at study entry:

* Male or female adult residents aged 18-40 years or children aged 1- 17 years who the investigator believes will comply with the requirements of the protocol (i.e. available for follow-up visits and specimen collection)
* For females of reproductive age, they must not be pregnant (as determined by verbal screening)
* Written informed consent obtained from subjects or their guardians, and written assent for children aged 12-17 years.
* Healthy subjects as determined by: medical history, physical examination, clinical judgement of the investigator.

Exclusion Criteria:

* Ongoing serious chronic disease
* Immunocompromising condition or therapy
* Diarrhea (3 or more loose stools within a 24-hour period) 6 weeks prior to enrollment
* one or two episodes of diarrhea lasting for more than 2 weeks in the past 6 months
* one or two episodes of abdominal pain lasting for more than 2 weeks in the past 6 months
* intake of any anti-diarrhoeal medicine in the past week
* abdominal pain or cramps, loss of appetite, nausea, general ill-feeling or vomiting in the past 24 hours
* acute disease one week prior to enrollment, with or without fever. Temperature > or = 38 degrees C (oral) or axillary temperature > or = 37.5 degrees C warrants deferral of the vaccination pending recovery of the subject
* receipt of antibiotics in past 14 days
* receipt of live or killed enteric vaccine in last month
* receipt of killed oral cholear vaccine

Ages: 1 Year to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2007-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects exhibiting 4-fold or greater rises in titers of serum vibriocidal antibodies, relative to baseline | 14 days after each dose of vaccine or placebo

SECONDARY OUTCOMES:
Geometric mean serum vibriocidal titers compared to baseline | 14 days after each dose
Proportion of subjects with any of the following adverse events: immediate reactions within 30 minutes after each dose and up to 3 days after each dose and serious adverse events occurring throughout the trial. | after dosing: 30 minutes to 3 days for adverse events, 28 days for serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Sujit K Bhattacharya, Principal Investigator — National Institute of Cholera and Enteric Diseases, India
Locations (1):
- National Institute of Cholera and Enteric Diseases, Kolkata, West Bengal, India

REFERENCES:
- [Result] Kanungo S, Paisley A, Lopez AL, Bhattacharya M, Manna B, Kim DR, Han SH, Attridge S, Carbis R, Rao R, Holmgren J, Clemens JD, Sur D. Immune responses following one and two doses of the reformulated, bivalent, killed, whole-cell, oral cholera vaccine among adults and children in Kolkata, India: a randomized, placebo-controlled trial. Vaccine. 2009 Nov 16;27(49):6887-93. doi: 10.1016/j.vaccine.2009.09.008. Epub 2009 Sep 15. PMID 19761838